CLINICAL TRIAL: NCT03806374
Title: Is it Possible to Replace Fentanyl by Non Narcotic Medication for Induction and Maintenance of Anesthesia in Minor Procedures?
Brief Title: Is it Possible to Replace Fentanyl in Anesthesia for Minor Procedures?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ayman Anis Metry, Assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ASUH9418
Record Dates: First submitted 2018-12-11; First posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Anesthesia
Keywords: fentanyl; lidocaine; ketamine; induction of anesthesia; intubation
MeSH Terms: interventions — Ketamine; Propofol; Fentanyl; cisatracurium; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fentanyl (Active Comparator): Administered propofol and fentanyl for induction.
  Interventions: Drug: Propofol; Drug: Fentanyl; Drug: Cisatracurium
- Ketamine and lidocaine (Active Comparator): Administered propofol, ketamine and lidocaine for induction.
  Interventions: Drug: Ketamine; Drug: Propofol; Drug: Cisatracurium; Drug: Lidocaine

INTERVENTIONS:
Drug: Ketamine — ketamine
  Arms: Ketamine and lidocaine
Drug: Propofol — propofol
Drug: Fentanyl — fentanyl
  Arms: Fentanyl
Drug: Cisatracurium — cisatracurium
Drug: Lidocaine — lidocaine
  Arms: Ketamine and lidocaine

SUMMARY:
To compare between fentanyl group and ketamine lidocaine group for induction of anesthesia as regards hemodynamics and smooth intubation.

DETAILED DESCRIPTION:
Two groups each with 60 patients Group I anesthesia initiated by propofol, fentanyl and cisatracurium. Group II anesthesia initiated by ketamine, lidocaine, propofol and cisatracurium.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II between
* Age between 18-55 years
* Undergoing minor surgical procedure less than an hour.

Exclusion Criteria:

* Patients with hypertension
* Patients with Ischemic heart diseases
* Patients with chronic renal or liver diseases

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
Intubation with less hemodynamic changes | 15 minutes after induction of anesthesia.
  changes in blood pressure with intubation
Smooth Maintenance of anesthesia | anesthesia time
  changes in blood pressure during anesthesia
less postoperative pain killers | 24 hours postoperative
  amount of pain killers used and timing
Intubation with less hemodynamic changes | Anesthesia time
  changes in pulse rate during anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No